CLINICAL TRIAL: NCT04981834
Title: The Effect of Vesicopexy on Urinary Continence and Quality of Life Following Robotic-Assisted Radical Prostatectomy: A Phase III Randomized Clinical Trial
Brief Title: Robot-Assisted Radical Prostatectomy With or Without Vesicopexy in Patients With Prostate Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual goal reached and suspended for analysis purposes.
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4P-21-1; NCI-2021-05989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-21-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2021-07-27; First posted 2021-07-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (radical prostatectomy, vesicopexy) (Experimental): Patients undergo standard RARP with anterior approach plus vesicopexy. Urethral catheters are removed 7-14 days following surgery at provider discretion.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy; Procedure: Vesicopexy
- Arm II (radical prostatectomy) (Active Comparator): Patients undergo standard RARP with anterior approach without vesicopexy. Urethral catheters are removed 7-14 days following surgery at provider discretion.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Radical Prostatectomy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Radical Prostatectomy — Undergo RARP
  Other Names: Prostatovesiculectomy
Procedure: Vesicopexy — Undergo vesicopexy
  Other Names: Cystopexy; Vesicofixation
  Arms: Arm I (radical prostatectomy, vesicopexy)

SUMMARY:
This phase III trial compares the effects of robot-assisted radical prostatectomy (RARP) with or without vesicopexy on urinary continence (a person's ability to control their bladder) and quality of life in patients with cancer of the prostate. RARP is the most adopted surgical approach for treatment of prostate cancer that has not spread to other places in the body (non-metastatic). Urinary incontinence (inability to control the bladder) is one of the most common complications of RARP, impacting patients' quality of life and psychological well-being. Different techniques have been proposed to improve urinary continence following RARP. Vesicopexy is one technique that restores the bladder to its normal position in the body after RARP. This study aims to evaluate whether RARP with vesicopexy may improve urinary continence and quality of life after surgery in prostate cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 3-month (+/- 3 weeks) urinary continence following RARP with or without vesicopexy.

SECONDARY OBJECTIVES:

I. To evaluate the 3-month (+/- 3 weeks) quality of life following RARP with or without vesicopexy.

II. To evaluate the 72-hour post-operative (postop) urinary continence following RARP with or without vesicopexy.

III. To evaluate the 1-month (+/- 1 week) postop urinary continence following RARP with or without vesicopexy.

IV. To evaluate sexual function at 3-month (+/- 3 weeks) following RARP with or without vesicopexy.

V. To evaluate the operative time in patients undergoing RARP with or without vesicopexy.

VI. To evaluate intraoperative complications in patients undergoing RARP with or without vesicopexy.

VII. To evaluate 90-day post-operative complications in patients undergoing RARP with or without vesicopexy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard RARP with anterior approach plus vesicopexy. Urethral catheters are removed 7-14 days following surgery at provider discretion.

ARM II: Patients undergo standard RARP with anterior approach without vesicopexy. Urethral catheters are removed 7-14 days following surgery at provider discretion.

After study completion, patients will be followed-up with at 24 hours, 1-month, and 3-months.

ELIGIBILITY:
Inclusion Criteria:

* Men with age > 18 years
* Prostate cancer patients undergoing RARP with anterior approach at University of Southern California (USC) urology
* Ability to understand and the willingness to sign a written informed consent
* Clinical stage < 4 and (M0) prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance score 0-1
* Pre-operative (op) urinary continence
* Negative history of pelvic radiation and/or previous local therapy for prostate cancer (i.e., radiation or focal therapy)

Exclusion Criteria:

* Any history of psychiatric, neurologic or cognitive disease
* Any history of neuropathic bladder
* Any drug or alcohol addiction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
3-month (+/- 3 weeks) urinary continence rate following RARP with or without vesicopexy | 3 months post-operative
  Defined continence as 0-1 safety pad usage. Use the "pictorial pad usage questionnaire."

SECONDARY OUTCOMES:
3-month (+/- 3 weeks) quality of life following surgery | 3 months post-operative
  Use the European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire (EORTC QLQ-PR25).
72-hour postop urinary continence following surgery | 72 hours post-operative
  Defined continence as 0-1 safety pad usage. Assessed with the "pictorial pad usage questionnaire."
1-month (+/- 1 week) post-operative urinary continence following surgery | 1 month post-operative
  Defined continence as 0-1 safety pad usage. Assessed with the "pictorial pad usage questionnaire."
Sexual function at 3-month (+/- 3 weeks) following surgery | 3 months post-operative
  Sexual Health Inventory for Men (SHIM) questionnaire is used for the evaluation of sexual function.
Operative time | Duration of operation
Intra-operative complications | Duration of operation
90-day post-operative complications | 90 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Djaladat, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States